CLINICAL TRIAL: NCT03560882
Title: A Pilot Trial of Atorvastatin in p53-Mutant and p53 Wild-Type Malignancies
Brief Title: A Pilot Trial of Atorvastatin in Tumor Protein 53 (p53) -Mutant and p53 Wild-Type Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joaquina Baranda (Other)
Responsible Party: Sponsor-Investigator, Joaquina Baranda, Associate Professor University of Kansas Cancer Center - Medical Oncology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2018-p53Atorva
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Malignant Disease; Solid Tumor; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Cancer; Relapsed Hematologic Malignancy
Keywords: atorvastatin; p53; tumor resection
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neoplasms; Hematologic Neoplasms | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atorvastatin (Experimental): Atorvastatin 80 milligrams (mg) per day, orally for 1 - 4 weeks before surgery (surgery not part of clinical trial)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin tablet, 80mg

SUMMARY:
This is a window-of-opportunity trial to determine if atorvastatin given for 1 to 4 weeks at a dose of 80 milligrams per day (mg/day) is sufficient to decrease the level of conformational mutant tumor protein 53 (p53) in malignant diseases (solid tumor and relapsed Acute Myeloid Leukemia (AML)).

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant to understand this study, and participant to sign a written informed consent. Legally authorized representative is not allowed to sign consent for participant.
* Participants with tumor protein 53 (TP53) immunohistochemistry (IHC)-positive tumors
* Participants whose screening IHC shows TP53-IHC-negative including wild type (WT) and null.
* Participants with histologic or cytologic confirmation of any malignant disease who are planning and eligible to undergo surgical resection. For participants with Solid Tumors Only
* Participants with previously treated acute myeloid leukemia (AML) are eligible if they relapse and are in between two treatment regimens
* No concurrent or recent (within 30 days) use of systemic therapy including chemotherapy, immunotherapy, hormonal therapy, cancer vaccine, or local therapy for the cancer.
* Formalin-fixed paraffin-embedded (FFPE) tumor tissue deemed adequate for IHC analysis and next generation sequencing (NGS) are required. Bone marrow aspirate tissue samples from participants with AML are required.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ and marrow function
* A negative urine or serum pregnancy test within 7 days before Day 1 dose of study medication, if female participant is of childbearing potential.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use two forms of adequate contraception (hormonal AND barrier method of birth control) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Current or anticipated use of other investigational agents while participating in this study.
* Pregnant or breast feeding.
* Diagnosis of squamous cell cancer of the oropharynx
* Previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast), unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period
* Prior use of statins in the past 30 days.
* History of rhabdomyolysis
* Active liver disease
* Participants who currently consume substantial quantities of alcohol (Male, more than 4 drinks a day, Female, more than 2 drinks a day)
* Concurrent use of drugs associated with myopathy
* Hypersensitivity to atorvastatin or any component of the formulation
* Untreated hypothyroidism
* Inability to comply with study and follow-up procedures as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in conformational mutant tumor protein 53 (p53) | baseline and up to 4 weeks
  Measured by immunohistochemistry (IHC) staining. Reported as overall percent difference in the level of conformation mutant p53.

SECONDARY OUTCOMES:
Change in Ki-67 (protein) | baseline and up to 4 weeks
  Measured by immunohistochemistry (IHC) staining. Reported as overall percent difference in the level of Ki-67 (also known as MKI67) in the conformation mutant p53 samples.
Change in caspase-3 | baseline and up to 4 weeks
  Measured by immunohistochemistry (IHC) staining. Reported as overall percent difference in the level of caspase-3 in the conformation mutant p53 samples.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquina Baranda, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (1):
- University of Kansas Cancer Center - CRC, Fairway, Kansas, United States

IPD SHARING:
Plan to Share IPD: No